CLINICAL TRIAL: NCT04396470
Title: Transcutaneous Vagus Nerve Stimulation in Children With Prader-Willi Syndrome
Brief Title: tVNS in Children With Prader-Willi Syndrome
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding received
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karen Parker, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 55936
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Prader-Willi Syndrome; Social Behavior
MeSH Terms: conditions — Prader-Willi Syndrome; Social Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tVNS treatment (Experimental)
  Interventions: Device: tVNS
- tVNS sham treatment (Sham Comparator)
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tVNS — Participants will be randomized to either the tVNS treatment condition or the sham tVNS (placebo) condition. An identical non-invasive tVNS device will be used in both groups. In the active condition, the device is placed on the external earlobe (tragus), which directly stimulates the vagus nerve. In the sham condition, the device is placed on the external earlobe, providing the same sensations as in the treatment condition, but no stimulation to the vagus nerve. Intervention period: Participants will use the device 1-hr per day for 12 weeks per manufacturer's instructions.

SUMMARY:
The purpose of the current project is to test the impact of transcutaneous vagus nerve stimulation (tVNS) on social ability in children with Prader-Willi Syndrome (PWS). Social ability and blood neuropeptides associated with social functioning will be measured before and after engagement in 12 weeks of tVNS therapy.

ELIGIBILITY:
Inclusion Criteria:

* (1) be between the ages of 8-14 years; (2) have a confirmed diagnosis of PWS by genetic testing; (3) be minimally verbal and able to sit at a table to complete cognitive and behavioral testing; (4) be willing to provide blood samples; and (5) be willing to engage in a 16-week study period (baseline to intervention follow-up).

Exclusion Criteria:

* (1) currently taking oxytocin and/or arginine vasopressin or related analogs and (2) have a DSM-5 diagnosis of any severe mental or behavioral disorder (e.g. schizophrenia, bipolar disorder, conduct or oppositional defiant disorder) that significantly impacts daily functioning.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, 2nd Edition (SRS-2) | pre-post 12 week intervention period
  Identifies the presence and severity of social impairments in child participants by parent report

IPD SHARING:
Plan to Share IPD: No